CLINICAL TRIAL: NCT04104529
Title: Establishment of a Clinico-biological Database in Patients Treated With Metabolic Radiotherapy in the Nuclear Medicine Department
Brief Title: Clinico-biological Database in Patients Treated With Metabolic Radiotherapy in the Nuclear Medicine Department
Acronym: BCB RIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2019-10 BRI
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Cancer; Prostate Cancer; Neuroendocrine Tumors
Keywords: thyroid cancer; prostate cancer; neuroendocrine tumors; nuclear medecine
MeSH Terms: conditions — Thyroid Neoplasms; Prostatic Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): Biological collection
  For all the patients include in the study :
  samples of blood samples collected before and during treatment. In parallel to this biological collection, standardized clinical data will be entered into a database
  Ancillary study :
  For metastatic thyroïd cancer and neuroendocrine tumor : anapath blocks of the initial diagnosis will be archived and dosimetric data will be collected for the cycle 1 For neuroendocrine tumor : blood sample additionnal will be realized at the cycle 1 (pre and post treatment)
  Interventions: Other: Biological collection; Other: tumor collection

INTERVENTIONS:
Other: Biological collection — The biological collection will also include samples of blood samples collected before and during treatment.
Other: tumor collection — Tumor collection (diagnosis) will be done for thyroid cancer and neuroencrine

SUMMARY:
Development of a clinico-biological database allowing the provision of clinical data and corresponding biological materials to the medical and scientific community.

DETAILED DESCRIPTION:
Targeted radionuclide therapy (TRT) aims at delivering ionizing radiation specifically to tumors for therapeutic purposes. Different types of radionuclides can be used to deliver the radiation: beta emitters less (Iodine-131, Lutecium-177), alpha (Radium-223) or Auger (Indium-111). They will target tumor cells either by natural tropism (iodine for thyroid cancer, for example) or by coupling them to a vector (antibody, peptide ...).

Patients with thyroid cancer, prostate cancer or neuroendocrine tumors who should benefit form TRT may be included in this project. The clinical-biological database will help better understanding of the radiobiological mechanisms of action of ionizing radiations on both normal tissues and tumor cells and the psycho-oncological mechanisms involved in patients treated with TRT (only for ICM's patients). The collected data will help treatment optimization.

To meet these demands, the research must then integrate databases creation open to researchers and the ongoing evaluation of the impact of projects on the health of cancer patients. Integrated research associated with quality biological research is the guarantee of medical progress. The multidisciplinary structure around collections of biological resources will enable the various actors to harmonize not only the collection but also the sharing of their data with a view to making them available for medico-scientific projects at a regional and national dimension. The Clinical Biological Database (BCB) should be used to identify and characterize new molecular markers for better diagnosis and / or treatment. It should also permit to optimize the collection of all this information, their integration and their transversal exploitation by different research disciplines (epidemiological, fundamental, translational, clinical).

An ancillary study "IMMUNORIV" is associated to BCB RIV : The specific research aim is, first, to determine whether immune cell (lymphocytes and macrophages) scoring and characterization in metastatic thyroid cancer and NET samples at diagnosis predict the response to TRT. Second, a high-throughput approach will be used to determine i) the immune cell profile in blood samples from patients with NET, before and after TRT initiation, and ii) its possible correlation with the response to TRT. Third, using imaging techniques the possible correlation will be evaluated between tumor uptake/absorbed dose and response to TRT.

By monitoring the immune response during TRT, the IMMUNORIV project will allow to identify immune response-related biomarkers that may be modulated to improve TRT effect.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ at 18 years old,
* Patient treated in the Nuclear Medicine Department for the treatment by metabolic radiotherapy,
* Patient treated as part of his treatment for:

  * thyroid cancer,
  * a neuroendocrine tumor or
  * prostate cancer.
* Patient having accepted the complementary blood sample,
* Patient having given his informed, written and express consent.

Exclusion Criteria:

* Patient not affiliated to a social security scheme,
* Subject under tutelage, curatorship or safeguard of justice,
* Patient in an emergency situation
* Patient whose regular monitoring is a priori impossible for psychological, family, social or geographical reasons,
* Pregnant and / or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who gave their consent to participate in the study | Until the study completion: 5 years
  The proportion of patients who consent to participate in the study among the screened patients

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DESHAYES, MD, Study Chair — Institut régional du Cancer Montpellier
Locations (4):
- France (4):
  - Hopital Haut Lévêque, Bordeaux, Aquitaine
  - Hôpital LaTimone, Marseille, Bouches Du Rhône
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Institut Universitaire du Cancer de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients
Supporting Information: Study Protocol

REFERENCES:
- [Background] Pouget JP, Lozza C, Deshayes E, Boudousq V, Navarro-Teulon I. Introduction to radiobiology of targeted radionuclide therapy. Front Med (Lausanne). 2015 Mar 17;2:12. doi: 10.3389/fmed.2015.00012. eCollection 2015. PMID 25853132
- [Background] Kumar C, Shetake N, Desai S, Kumar A, Samuel G, Pandey BN. Relevance of radiobiological concepts in radionuclide therapy of cancer. Int J Radiat Biol. 2016;92(4):173-86. doi: 10.3109/09553002.2016.1144944. Epub 2016 Feb 26. PMID 26917443
- [Background] Gudkov SV, Shilyagina NY, Vodeneev VA, Zvyagin AV. Targeted Radionuclide Therapy of Human Tumors. Int J Mol Sci. 2015 Dec 28;17(1):33. doi: 10.3390/ijms17010033. PMID 26729091
- [Background] Schlumberger M, Catargi B, Borget I, Deandreis D, Zerdoud S, Bridji B, Bardet S, Leenhardt L, Bastie D, Schvartz C, Vera P, Morel O, Benisvy D, Bournaud C, Bonichon F, Dejax C, Toubert ME, Leboulleux S, Ricard M, Benhamou E; Tumeurs de la Thyroide Refractaires Network for the Essai Stimulation Ablation Equivalence Trial. Strategies of radioiodine ablation in patients with low-risk thyroid cancer. N Engl J Med. 2012 May 3;366(18):1663-73. doi: 10.1056/NEJMoa1108586. PMID 22551127
- [Background] Dizdarevic S, Tulchinsky M, McCready VR, Mihailovic J, Vinjamuri S, Buscombe JR, Lee ST, Frangos S, Sathekge M, Siraj Q, Choudhury P, Bom H, Franceschi M, Ugrinska A, Paez D, Hussain R, Mailman J, Luster M, Virgolini I; WARMTH Thyroid Group. The World Association of Radiopharmaceutical and Molecular Therapy position statement on the initial radioiodine therapy for differentiated thyroid carcinoma. World J Nucl Med. 2019 Apr-Jun;18(2):123-126. doi: 10.4103/wjnm.WJNM_117_18. No abstract available. PMID 31040741
- [Background] Strosberg J, El-Haddad G, Wolin E, Hendifar A, Yao J, Chasen B, Mittra E, Kunz PL, Kulke MH, Jacene H, Bushnell D, O'Dorisio TM, Baum RP, Kulkarni HR, Caplin M, Lebtahi R, Hobday T, Delpassand E, Van Cutsem E, Benson A, Srirajaskanthan R, Pavel M, Mora J, Berlin J, Grande E, Reed N, Seregni E, Oberg K, Lopera Sierra M, Santoro P, Thevenet T, Erion JL, Ruszniewski P, Kwekkeboom D, Krenning E; NETTER-1 Trial Investigators. Phase 3 Trial of 177Lu-Dotatate for Midgut Neuroendocrine Tumors. N Engl J Med. 2017 Jan 12;376(2):125-135. doi: 10.1056/NEJMoa1607427. PMID 28076709
- [Background] Strosberg JR, Halfdanarson TR, Bellizzi AM, Chan JA, Dillon JS, Heaney AP, Kunz PL, O'Dorisio TM, Salem R, Segelov E, Howe JR, Pommier RF, Brendtro K, Bashir MA, Singh S, Soulen MC, Tang L, Zacks JS, Yao JC, Bergsland EK. The North American Neuroendocrine Tumor Society Consensus Guidelines for Surveillance and Medical Management of Midgut Neuroendocrine Tumors. Pancreas. 2017 Jul;46(6):707-714. doi: 10.1097/MPA.0000000000000850. PMID 28609356
- [Background] Parker C, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Seke M, Widmark A, Johannessen DC, Hoskin P, Bottomley D, James ND, Solberg A, Syndikus I, Kliment J, Wedel S, Boehmer S, Dall'Oglio M, Franzen L, Coleman R, Vogelzang NJ, O'Bryan-Tear CG, Staudacher K, Garcia-Vargas J, Shan M, Bruland OS, Sartor O; ALSYMPCA Investigators. Alpha emitter radium-223 and survival in metastatic prostate cancer. N Engl J Med. 2013 Jul 18;369(3):213-23. doi: 10.1056/NEJMoa1213755. PMID 23863050
- [Background] Domenech A, Notta P, Benitez A, Ramal D, Rodriguez-Bel L, Massuet C, Martin-Comin J. [Evaluation of the anxiety state in patients receiving radioiodine treatment or who undergo a sentinel lymph node examination in the Nuclear Medicine Department]. Rev Esp Med Nucl. 2010 Mar-Apr;29(2):63-72. doi: 10.1016/j.remn.2009.12.009. Epub 2010 Feb 18. Spanish. PMID 20167394
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Background] Arrieta O, Angulo LP, Nunez-Valencia C, Dorantes-Gallareta Y, Macedo EO, Martinez-Lopez D, Alvarado S, Corona-Cruz JF, Onate-Ocana LF. Association of depression and anxiety on quality of life, treatment adherence, and prognosis in patients with advanced non-small cell lung cancer. Ann Surg Oncol. 2013 Jun;20(6):1941-8. doi: 10.1245/s10434-012-2793-5. Epub 2012 Dec 22. PMID 23263699
- [Background] Barbus E, Pestean C, Larg MI, Gabora K, Bonci EA, Badulescu C, Piciu A. Psychological impact of 131I radioprotection measures on thyroid cancer patients. Clujul Med. 2018 Oct;91(4):441-447. doi: 10.15386/cjmed-1042. Epub 2018 Oct 30. PMID 30564021
- [Background] De Vincentis G, Frantellizzi V, Follacchio GA, Farcomeni A, Pani A, Samaritani R, Schinzari G, Santini D, Cortesi E. No evidence of association between psychological distress and pain relief in patients with bone metastases from castration-resistant prostate cancer treated with 223Radium. Eur J Cancer Care (Engl). 2019 Sep;28(5):e13112. doi: 10.1111/ecc.13112. Epub 2019 May 31. PMID 31148330
- [Background] Strosberg J, Wolin E, Chasen B, Kulke M, Bushnell D, Caplin M, Baum RP, Kunz P, Hobday T, Hendifar A, Oberg K, Sierra ML, Thevenet T, Margalet I, Ruszniewski P, Krenning E; NETTER-1 Study Group. Health-Related Quality of Life in Patients With Progressive Midgut Neuroendocrine Tumors Treated With 177Lu-Dotatate in the Phase III NETTER-1 Trial. J Clin Oncol. 2018 Sep 1;36(25):2578-2584. doi: 10.1200/JCO.2018.78.5865. Epub 2018 Jun 7. PMID 29878866
- [Background] Prieto JM, Blanch J, Atala J, Carreras E, Rovira M, Cirera E, Gasto C. Psychiatric morbidity and impact on hospital length of stay among hematologic cancer patients receiving stem-cell transplantation. J Clin Oncol. 2002 Apr 1;20(7):1907-17. doi: 10.1200/JCO.2002.07.101. PMID 11919251
- [Background] Kim Y, Spillers RL. Quality of life of family caregivers at 2 years after a relative's cancer diagnosis. Psychooncology. 2010 Apr;19(4):431-40. doi: 10.1002/pon.1576. PMID 19399773
- [Background] Lloyd-Williams M, Dennis M, Taylor F. A prospective study to determine the association between physical symptoms and depression in patients with advanced cancer. Palliat Med. 2004 Sep;18(6):558-63. doi: 10.1191/0269216304pm923oa. PMID 15453627
- [Background] Satin JR, Linden W, Phillips MJ. Depression as a predictor of disease progression and mortality in cancer patients: a meta-analysis. Cancer. 2009 Nov 15;115(22):5349-61. doi: 10.1002/cncr.24561. PMID 19753617
- [Background] Pinquart M, Duberstein PR. Depression and cancer mortality: a meta-analysis. Psychol Med. 2010 Nov;40(11):1797-810. doi: 10.1017/S0033291709992285. Epub 2010 Jan 20. PMID 20085667
- [Background] Schouten B, Avau B, Bekkering GTE, Vankrunkelsven P, Mebis J, Hellings J, Van Hecke A. Systematic screening and assessment of psychosocial well-being and care needs of people with cancer. Cochrane Database Syst Rev. 2019 Mar 26;3(3):CD012387. doi: 10.1002/14651858.CD012387.pub2. PMID 30909317
- [Background] Pirl WF, Fann JR, Greer JA, Braun I, Deshields T, Fulcher C, Harvey E, Holland J, Kennedy V, Lazenby M, Wagner L, Underhill M, Walker DK, Zabora J, Zebrack B, Bardwell WA. Recommendations for the implementation of distress screening programs in cancer centers: report from the American Psychosocial Oncology Society (APOS), Association of Oncology Social Work (AOSW), and Oncology Nursing Society (ONS) joint task force. Cancer. 2014 Oct 1;120(19):2946-54. doi: 10.1002/cncr.28750. Epub 2014 May 2. PMID 24798107
- [Background] Wu HX, Zhong H, Xu YD, Xu CP, Zhang Y, Zhang W. Psychological and behavioral intervention improves the quality of life and mental health of patients suffering from differentiated thyroid cancer treated with postoperative radioactive iodine-131. Neuropsychiatr Dis Treat. 2016 May 2;12:1055-60. doi: 10.2147/NDT.S105460. eCollection 2016. PMID 27194911
- [Background] Dolbeault S, Bredart A, Mignot V, Hardy P, Gauvain-Piquard A, Mandereau L, Asselain B, Medioni J. Screening for psychological distress in two French cancer centers: feasibility and performance of the adapted distress thermometer. Palliat Support Care. 2008 Jun;6(2):107-17. doi: 10.1017/S1478951508000187. PMID 18501045
- [Background] Shou J, Zhang Z, Lai Y, Chen Z, Huang J. Worse outcome in breast cancer with higher tumor-infiltrating FOXP3+ Tregs : a systematic review and meta-analysis. BMC Cancer. 2016 Aug 26;16(1):687. doi: 10.1186/s12885-016-2732-0. PMID 27566250
- [Background] Constanzo J, Parach A, David T, Karam J, Bruchertseifer F, Morgenstern A, Jarlier M, Bardies M, Deshayes E, Gudin-de-Vallerin A, Boissiere-Michot F, Lopez-Crapez E, Pouget JP. MHC-I-Driven Antitumor Immunity Counterbalances Low Absorbed Doses of Radiopharmaceutical Therapy. J Nucl Med. 2025 May 1;66(5):785-792. doi: 10.2967/jnumed.124.268857. PMID 40015918